CLINICAL TRIAL: NCT01283386
Title: Prospective Randomized Study to Compare Efficacy and Safety of RFC-Lite (Rituximab, Fludarabine, Cyclophosphamide) Regimen With LR (Rituximab, Chlorambucil) as a First-Line Therapy in Patients With B-Cell Chronic Lymphocytic Leukemia and Unfavorable Somatic Status
Brief Title: A Study to Compare Mabthera (Rituximab), Fludarabine and Cyclophosphamide to Mabthera and Chlorambucil in Participants With Chronic Lymphocytic Leukemia and Unfavorable Somatic Status
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25137
Record Dates: First submitted 2011-01-18; First posted 2011-01-26 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; Cyclophosphamide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCR-lite (Experimental): Rituximab, fludarabine, and cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab
- LR Therapy (Active Comparator): Rituximab and chlorambucile
  Interventions: Drug: Chlorambucil; Drug: Rituximab

INTERVENTIONS:
Drug: Chlorambucil — 10 mg/m^2 orally on Days 1-7 of each 28-day cycle for 6 cycles
  Arms: LR Therapy
Drug: Cyclophosphamide — 150 mg/m^2 IV or orally on Days 1-3 of each 28-day cycle for 6 cycles
  Arms: FCR-lite
Drug: Fludarabine — 20 mg/m^2 IV or 32 mg/m2 orally Days 1-3 of each 28-day cycle for 6 cycles
  Arms: FCR-lite
Drug: Rituximab — 375 mg/m2 IV on Day 1 of Cycle 1; 500 mg/m2 IV on Day 1 of Cycles 2-6 (28-day cycles)
  Other Names: MabThera

SUMMARY:
This multi-center, randomized study compared the efficacy and safety of MabThera (rituximab) in combination with either fludarabine and cyclophosphamide or with chlorambucil in participants with previously untreated B-cell chronic lymphocytic leukemia and unfavorable somatic status. Participants were randomized to receive Mabthera (375 mg/m2 intravenously [IV] Day 1 of Cycle 1, 500 mg/m2 IV Day 1 Cycles 2-6) with either fludarabine (20 mg/m2 IV or 32 mg/m2 orally Days 1-3) and cyclophosphamide (150 mg/m2 IV or orally Days 1-3) or with chlorambucil (10 mg/m2 orally Days 1-7) for 6 cycles of 28 days. Anticipated time on study treatment was 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 60-70 or >70 years of age
* Cumulative Illness Rating Scale (CIRS) comorbidity score >/=7 if patient is 60-70 years old
* Previously untreated B-cell chronic lymphocytic leukemia
* Binet stage B, C or A with progression
* ECOG performance status 0-2

Exclusion Criteria:

* Small-cell lymphoma
* Autoimmune hemolytic anemia
* Concomitant malignant disease during enrollment, except for basal cell carcinoma of the skin
* Chemotherapy for concomitant malignant disease within 12 months prior to study enrollment
* Richter's syndrome

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Russia (8):
  - The order of Honour pin Irkutsk regional clinical hospital; Hematology Department, Irkutsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - City Clinical Botkin's Hospital; City Hematological Center, Moscow
  - Saint-Petersburg SHI City Clinical Hospital #31, Saint Petersburg
  - City Clinical Hospital #15; Hematology department, Saint Petersburg
  - GUZ Tula Regioanal Clinical Hospital; Hematology, Tula
  - Republican clinical hospital named after G.G. Kuvatov, Ufa

RESULTS

PARTICIPANT FLOW:
Groups:
- FCR-lite: Rituximab 375 milligrams per square meter (mg/m^2) intravenously (IV) on Day 1 of Cycle 1 (one cycle = 28 days), then 500 mg/m^2 IV on Day 1 of each subsequent cycle for 6 cycles. When fludarabine / cyclophosphamide IV administered: fludarabine 20 mg/m^2 IV on Days 1-3; cyclophosphamide 150 mg/m^2 IV on Days 1-3. When fludarabine / cyclophosphamide orally administered: fludarabine 32 mg/m^2 orally on Days 1-3; cyclophosphamide 150 mg/m^2 orally on Days 1-3 for 6 cycles (28 days each).
- LR Therapy: Rituximab 375 mg/m^2 IV on Day 1 of Cycle 1, then 500 mg/m^2 IV on Day 1 of each subsequent cycle for 6 cycles. Chlorambucile 10 mg/m^2 orally on Days 1-7 for 6 cycles.
Period: Overall Study
Arm/Group | FCR-lite | LR Therapy
Started | 10 | 16
Completed | 2 | 4
Not Completed | 8 | 12
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Relapse of underlying disease | 1 | 3
Not completed — Progression of underlying disease | 2 | 7
Not completed — Reason not specified | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FCR-lite | LR Therapy | Total
Number analyzed (Participants) | 10 | 16 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (7.09) | 68.6 (4.95) | 68.6 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission
Description: Complete remission was defined as the disappearance of all signs of disease.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure at the end of therapy.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 7 | 16
percentage of participants | 42.9 | 18.8

2. Primary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure at the end of therapy.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 7 | 16
percentage of participants | 0 | 6.3

3. Primary Outcome: Percentage of Participants With Stable Disease
Description: Stable disease was defined as not meeting the criteria for partial remission or disease progression
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure at the end of therapy.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 7 | 16
percentage of participants | 14.3 | 18.8

4. Primary Outcome: Percentage of Participants With Partial Remission
Description: Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure at the end of therapy.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 7 | 16
percentage of participants | 42.9 | 56.3

5. Primary Outcome: Duration of Response
Description: Duration of Response was defined as the time period from the last day of study treatment to the day when disease progression occurred in participants who previously had complete or partial remission. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen. Complete remission was defined as the disappearance of all signs of disease. Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who had disease progression after response to therapy.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 5 | 12
days | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events. | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events.

6. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time period from the first day of study treatment to the day when disease progression occurred. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who had disease progression at the end of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 8 | 16
days | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events. | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events.

7. Primary Outcome: Event-free Survival
Description: Event-free survival was defined as the time period from the first day of study treatment to occurrence of any of the following events: appearance of disease progression or relapse; prescription of a new treatment for disease relapse; death caused by B-cell chronic lymphocytic leukemia (B-CLL); or complications from B-CLL or therapy. Relapse was defined as disease progression in participants with complete or partial remission lasting at least 6 months after treatment completion. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen. Complete remission was defined as the disappearance of all signs of disease. Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who had an event of disease progression, relapse, or death.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 9 | 16
days | 679 [14.00 to NA] — 95% upper confidence interval limit was not calculable due to the low numbers of participants with events. | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events.

8. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time period from the first day of study treatment to participant death.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who died.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 10 | 16
days | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events. | NA [NA to NA] — Median and 95% lower and upper confidence interval limits were not calculable due to the low numbers of participants with events.

9. Primary Outcome: Percentage of Participants With Phenotypic Remission
Description: Phenotypic remission was considered achieved if a participant had a negative test for minimal residual disease. A negative test for minimal residual disease was defined as tumor cells ≤0.01% of the total number of peripheral leukocytes.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 8 | 10
percentage of participants | 25.0 | 30.0

10. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs
Description: An AE was defined as any unfavorable medical occurrence in a participant receiving a study drug, regardless of relationship the study drug. An AE was considered serious if it met any of the following criteria: was fatal or life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was clinically significant and/or required an intervention to prevent any of the listed criteria.
Time Frame: Up to approximately 5 years
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | FCR-lite | LR Therapy
Number analyzed (Participants) | 10 | 16
percentage of participants
  Non-serious AEs | 80.00 | 56.25
  Serious AEs | 20.00 | 18.75

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Arm/Group | FCR-lite | LR Therapy
Serious Adverse Events (participants affected / at risk) | 2/10 | 3/16
Other Adverse Events (participants affected / at risk) | 8/10 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FCR-lite (N=10) | LR Therapy (N=16)
Death (General disorders) | 2 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute myocardial infarction (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FCR-lite (N=10) | LR Therapy (N=16)
Neutrophil count decreased (Investigations) | 2 | 2
White blood cell count decreased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Glomerular filtration rate (Investigations) | 1 | 0
Urea urine increased (Investigations) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hyperglycaemia (Endocrine disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Chills (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.